CLINICAL TRIAL: NCT06164418
Title: Comparative Evaluation of Class V Restorations: 2-Year Randomized Double-Blind Trial Comparing Ion-Releasing Materials and Resin Composite
Brief Title: Comparative Evaluation of Class V Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hoda saleh, Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01011023 CD
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Secondary Caries; Dental Restoration Failure of Marginal Integrity

STUDY DESIGN:
Intervention Model Description: Each patient will receive one restoration in a posterior tooth on any side randomly selected from the 4 tested restorative systems groups, all materials will be used according to manufacturers' instructions
Who Masked: Participant, Investigator
Masking Description: Double (Participant and Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- a nanohybrid resin composite material with a universal adhesive (Placebo Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Procedure: Dental restoration
- a nanohybrid resin composite material with a fluoride-releasing universal adhesive (Active Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Procedure: Dental restoration
- ion-releasing restorative material with a universal adhesive (Placebo Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Procedure: Dental restoration
- ion-releasing restorative material with a fluoride-releasing universal adhesive (Active Comparator): Each patient will randomly receive one cervical restoration with one of the tested restorative systems
  Interventions: Procedure: Dental restoration

INTERVENTIONS:
Procedure: Dental restoration — Each patient will receive a cervical restoration using the corresponding group adhesive and restorative material

SUMMARY:
To evaluate and compare the 2-year clinical performance of Class V restorations using various restorative systems with ion-releasing and non-ion-releasing composites, utilizing fluoride-free and fluoride-releasing universal adhesives for bonding

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a double-blinded randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation. The trial will follow a parallel design. A total of one hundred adult patients, who are seeking dental treatment, will be enrolled in the study. The participants will be recruited from the Operative Department clinic at the Faculty of Dentistry, University of Mansoura. The study will focus on one hundred Class V restorations.

No active advertisement will be used for participant recruitment, and instead, a convenience sample will be formed. Prior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The study is scheduled to be conducted from November 2023 to November 2025. The form and protocol of the study will be approved by Mansoura University's ethics committee before initiation.

To determine the appropriate sample size, previous studies examining the clinical success rate of posterior class V restorations restored with ion-releasing materials were considered. These studies reported a 100% success rate at a two-year follow-up. Based on various parameters, including a significance level of 5%, a test power of 80%, and an equivalence limit of 15%, the sample size was calculated. Considering a potential dropout rate of 20%, a sample size of 100 subjects was determined to be suitable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one primary cervical caries on the buccal surface of any of their upper or lower posterior teeth. The cervical lesions must have an enamel margin occlusally and a cervical dentin margin
* Patients must have a good oral hygiene;
* Patients with tooth gives a positive response to testing with an electric pulp tester
* Patients with normal and full occlusion,
* Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

- High caries risk patients with extremely poor oral hygiene,

* Patients involved in orthodontic treatment or periodontal surgery,
* Patients with periodontally involved teeth (chronic periodontitis)
* Patients with heavy bruxism habits and clenching

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of aesthetic, functional and biological properties for each group | 2 years after restoration
  Percentage of aesthetic, functional and biological properties that will be clinically assessed using World Dental Federation parameters for each restorative system group

CONTACTS AND LOCATIONS:
Overall Officials: Hoda S Ismail, Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt
Locations (1):
- Hoda Saleh Ismail, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 Months for 2 years
Access Criteria: for anyone